CLINICAL TRIAL: NCT04704375
Title: Effects of Osteopathic Manipulative Treatment (OMT) and Bio Electro-Magnetic Regulation (BEMER) Therapy on Low Back Pain in Adults.
Brief Title: Effects of Osteopathic Manipulative Treatment and Bio Electro-Magnetic Regulation Therapy on Low Back Pain in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Santiago Lorenzo, PhD, Professor of Physiology, Lake Erie College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-154
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Musculoskeletal Pain
Keywords: OMM; BEMER
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Therapeutics; Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Bio Electro-Magnetic Regulation (BEMER) Therapy (Experimental): Subjects in the BEMER group received treatment 5 times per week for a period of 3 weeks.
  Interventions: Device: Bio Electro-Magnetic Regulation (BEMER) Therapy
- OMT (Osteopathic Manipulative Treatment) (Active Comparator): Each subject in the OMT group received treatment 3 times per week for a period of 3 weeks.
  Interventions: Procedure: OMT (osteopathic manipulative treatment)
- BEMER + OMT (Experimental): Each subject in the BEMER + OMT group received treatment 3 times per week for a period of 3 weeks.
  Interventions: Device: Bio Electro-Magnetic Regulation (BEMER) Therapy; Procedure: OMT (osteopathic manipulative treatment)
- Control (Sham Comparator): Finally, subjects in the Placebo group will receive the light touch and BEMER sham treatments at same intervals as the corresponding experimental groups.
  Interventions: Procedure: Light touch

INTERVENTIONS:
Device: Bio Electro-Magnetic Regulation (BEMER) Therapy — BEMER is a therapeutic modality that deploys a biorhythmically defined stimulus through Pulsed Electromagnetic Field (PEMF). This stimulus has a targeted effect on the microvasculature, and the primary effect is an improvement in tissue microcirculation. The positive effects of vasomotion on the microcirculation has been shown to result in significant increases in arteriovenous oxygen difference, number of open capillaries, arteriolar and venular flow volume, and flow rate of red blood cells in the microvasculature. Therefore, BEMER can potentially be used in the treatment of LBP by improving microcirculation in muscular tissue.
  Arms: BEMER + OMT; Bio Electro-Magnetic Regulation (BEMER) Therapy
Procedure: OMT (osteopathic manipulative treatment) — i. OMT Myofascial release (MFR), soft tissue (ST) release, muscle energy (ME), counterstrain (CS), and balanced ligamentous tension (BLT) technique.
  Arms: BEMER + OMT; OMT (Osteopathic Manipulative Treatment)
Procedure: Light touch — Treaters will place their hands lightly on the subject's lumbar paraspinal muscles in the supine and prone positions in the same area as where one would place your hands for lumbar MFR technique for the same amount of time as it would take to perform MFR in this area (approximately 5 minutes). However, no lifting or action will be done. In addition, the subject will lie down on the BEMER mat (as they would do during a BEMER session), but the device will not be activated.
  Arms: Control

SUMMARY:
It is clear that low back pain (LBP) is a major challenge in our society, which can lead to severe disability in many individuals. Although there are several different treatments and approaches to help individuals with LBP, the number affected by this condition has been steadily increasing.

OMT has been shown to be helpful in the treatment of LBP. In fact, the use of OMT has been shown to increase mobility of the lumbar myofascial tissues, visceral motion and decrease pain in patients with LBP. Bio Electro-Magnetic Regulation (BEMER) Therapy is a therapeutic modality that deploys a biorhythmically defined stimulus through a Pulsed Electromagnetic Field (PEMF), which leads to an increase in blood flow. The positive effects of BEMER on the circulation has been shown to result in significant increases in arteriovenous oxygen difference, number of open capillaries, arteriolar and venular flow volume, and flow rate of red blood cells in the microvasculature. Therefore, BEMER can potentially be used in the treatment of LBP by improving microcirculation in muscular tissue. In fact, BEMER with physiotherapy showed reductions in pain and fatigue acutely in patients with chronic low back pain. A systemic review of randomized controlled trials that investigated whether PEMF was effective in low back pain showed there was decrease in pain intensity and improved functionality in individuals with different low back pain conditions.

Therefore, it is plausible that the combination of OMT and BEMER therapy may help increase circulation to myofascial structures that influence low back restriction and pain. The purpose of this study is to investigate the individual and combined effects of OMT and BEMER therapy on low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) has become a major challenge in our society and has a relatively high incidence and prevalence. Moreover, LBP currently affects people of all ages and is a leading contributor to disease burden worldwide [6]. Individuals affected by LBP may experience this discomfort and associated disability for several months, and a proportion may remain severely disabled. For nearly all people with low back pain, it is not possible to identify a specific nociceptive cause. Most people with new episodes of LBP may recover quickly; however, recurrence is common and in many cases, LBP becomes persistent and disabling.

Despite the overabundance of treatments and approaches devoted to LBP, this back related disability and the number of individuals affected have steadily been increasing. During the past three decades, changes have been made to key recommendations in national clinical practice guidelines. In fact, currently there is a bigger emphasis placed on self-management, physical and psychological therapies, and some forms of complementary medicine (such as spinal manipulation, massage, acupuncture), and less emphasis on pharmacological and surgical treatments.

Despite multiple clinical guidelines providing similar recommendations for managing low back pain, a substantial gap between evidence and practice exists. Osteopathic manipulative treatment (OMT) is a distinctive modality used by osteopathic physicians to complement conventional management of LBP. There is considerable variability in OMT approaches when treating for LBP. Furthermore, osteopathic physicians combine conventional and complementary treatments when caring for patients with LBP. This increased variability in the approach to care for LBP patients requires more empirical data to determine the best approaches to treat LBP. Franke et al. conducted a meta-analysis that investigated the effect of OMT in LBP. The authors reported that some studies observed significant effect of OMT on pain, whereas other reported either a non-significant effect, or an effect in favor of the control treatment. It is clear that more research to better describe the effects of OMT on LBP is warranted.

OMT is the application of hands-on forces to help improve physiologic function and/or support homeostasis that has been negatively altered by somatic dysfunction, which is an impairment of function of any area of the body system. These impairments can occur at the muscles, fascia, bones, joints, ligaments, vasculature, lymphatics and nerves. When somatic dysfunction is diagnosed, using an osteopaths' manual palpatory skills, it is treated with OMT. In general, OMT techniques can be classified as direct or indirect. Direct techniques such as muscle energy (ME), high velocity low amplitude (HVLA), soft tissue (ST), and myofascial release (MFR) engage the restrictive barrier and use a specifically applied force to correct the somatic dysfunction [21]. Indirect techniques such as MFR, counterstrain (CS), balanced ligamentous tension (BLT) disengage from the restrictive barrier and the affected body part is moved into its freedom of motion.

The etiology of low back pain is varied from visceral causes, to a lack of adequate blood flow to the muscles and musculoskeletal imbalance. Inadequate blood supply and/or inadequate oxygen consumption can influence muscle pain. The role of OMT is thought to primarily address the musculoskeletal component of back pain, which may help improve muscle blood flow. Two of the primary goals of treatment with osteopathic techniques are to restore mobility and decrease pain. Using trained palpatory skills to diagnose alterations in the fascial connections within the body, it is proposed that OMT techniques can help alleviate these alterations in the body that may lead to musculoskeletal disorders such as low back pain. Many studies that use OMT as the intervention to reduce low back pain, utilize a combination of direct and indirect techniques. The use of myofascial release technique has been shown to increase mobility of the lumbar myofascial tissues, visceral motion and decrease pain in patients with non-specific low back pain using ultrasound diagnostics.

One very promising alternative approach for the treatment of LBP is the use of Bio Electro-Magnetic Regulation (BEMER) Therapy. BEMER is a therapeutic modality that deploys a biorhythmically defined stimulus through a Pulsed Electromagnetic Field (PEMF). This stimulus has a targeted effect on the microvasculature, and the primary effect is an improvement in tissue microcirculation. The positive effects of vasomotion on the microcirculation has been shown to result in significant increases in arteriovenous oxygen difference, number of open capillaries, arteriolar and venular flow volume, and flow rate of red blood cells in the microvasculature. Therefore, BEMER can potentially be used in the treatment of LBP by improving microcirculation in muscular tissue.

Though OMT has been shown to be effective clinically for patients in decreasing pain, little is known behind the specific mechanisms of action. It is believed all osteopathic techniques use the concepts of fascial connectivity throughout the body and therefore can help increase circulation and lymphatic flow. In one study, the use of OMT helped decrease autonomic and neuroendocrine markers in response to mental stress. In modeled studies, OMT modalities like MFR and CS showed possible effects in modifying cytokine secretion, improving wound healing, and modifying muscle contraction. These effects were shown to sometimes reverse repetitive muscle strain in the tissues. It is postulated that these strains may represent the phenomenon of somatic dysfunction. Another study showed improvement in lower extremity blood pressure, cell mass, intracellular water, basal metabolism, venous velocity, skin temperature, pain, and quality of life post MFR and physical therapy for post-menopausal women with venous insufficiency. As discussed previously, BEMER therapy has been shown to increase microcirculation. BEMER with physiotherapy showed reductions in pain and fatigue acutely in patients with chronic low back pain. A systemic review of randomized controlled trials that investigated whether PEMF was effective in low back pain showed there was decrease in pain intensity and improved functionality in individuals with different low back pain conditions [4]. Therefore the results from these studies suggest that the combination of OMT and BEMER therapy can potentially help increase circulation to myofascial structures that influence low back restriction and pain.

ELIGIBILITY:
Inclusion Criteria:

* LECOM-Bradenton faculty, staff and Students currently enrolled in LECOM-Bradenton's osteopathic medical program, pharmacy program, dental program, and master's program
* Currently experiencing low back pain.

Exclusion Criteria:

* Unable to provide informed consent
* Currently pregnant
* Medical history of current psychiatric conditions
* Skin disorders or open wounds precluding skin contact
* Fasciitis of fascial tears
* Myositis
* Neurological symptoms such as numbness, tingling, weakness in lower extremities
* Neoplasia
* Cancer
* Bone fracture, osteomyelitis, or osteoporosis,
* Coagulation problem
* Deep vein thrombosis
* Adrenal diseases/syndromes,
* Acute upper or lower respiratory infection
* Immunosuppressive syndromes
* Radiation or chemotherapy within the past 3 years
* Lupus
* Osteopenia
* Congestive heart failure
* BMI greater than 30
* Any other autoimmune disease not stated above
* Medication changes within the last 4 weeks
* Asthma exacerbations within the last 4 weeks
* Immunosuppressive therapy as a consequence of organ transplantation,
* Immunosuppressive therapy as a consequence of allogeneic cellular transplantations or bone marrow stem cell transplantation
* Other conditions often requiring immunosuppressive therapy, anticoagulant therapy, or known sensitivity to the carotid sinus reflex.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Lorenzo, PhD, Principal Investigator — Lake Erie College of Osteopathic Medicine
Locations (1):
- LECOM-Bradenton, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BEMER: Subjects in the BEMER group received treatment 5 times per week for a period of 3 weeks.
  Bio Electro-Magnetic Regulation (BEMER) Therapy: BEMER is a therapeutic modality that deploys a biorhythmically defined stimulus through Pulsed Electromagnetic Field (PEMF). This stimulus has a targeted effect on the microvasculature, and the primary effect is an improvement in tissue microcirculation. The positive effects of vasomotion on the microcirculation has been shown to result in significant increases in arteriovenous oxygen difference, number of open capillaries, arteriolar and venular flow volume, and flow rate of red blood cells in the microvasculature. Therefore, BEMER can potentially be used in the treatment of LBP by improving microcirculation in muscular tissue.
Period: Overall Study
Arm/Group | BEMER | OMT (Osteopathic Manipulative Treatment) | BEMER + OMT | Control
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BEMER | OMT (Osteopathic Manipulative Treatment) | BEMER + OMT | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 6 | 21
  Male | 6 | 5 | 4 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 10 | 10 | 40
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Visual Analog Scale [Mean (Standard Deviation); unit: units on a scale] — Scale range (0-100) to determine level of pain (0:no pain, 100: the most pain ever experienced)
  units on a scale | 44.5 (20.6) | 32.1 (25.2) | 38.2 (26.8) | 34.1 (26.0) | 37.2 (24.7)

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain Rating Visual Analog Scale
Description: Assessed by questionnaire rating, compared with pre-intervention rating
  Visual Analog Scale (VAS). Score ranges 0-100. Minimum score=0 (no pain), Maximum score=100 (worst pain ever felt). Lower scores is better as it reflect lower pain
Time Frame: Within 1 week of completion of 3-week intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMER | OMT (Osteopathic Manipulative Treatment) | BEMER + OMT | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 44.5 (20.6) | 32.1 (25.2) | 38.2 (26.8) | 34.1 (26)

2. Primary Outcome: Low Back Pain Rating Oswestry Low Back Pain Questionnaire
Description: Assessed by questionnaire rating, compared with pre-intervention rating
  Oswestry low back pain questionnaire: Scores range 0-50. 0-4 indicating no disability; 5-14 indicating minimal disability; 15-24 moderate disability; 25-34 severe disability; 35-50 complete disability. Lower scores is better as it reflect lower pain
Time Frame: Within 1 week of completion of 3-week intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMER | OMT (Osteopathic Manipulative Treatment) | BEMER + OMT | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 14.8 (10.8) | 14.4 (12.1) | 11.2 (10.8) | 10.8 (9.0)

3. Primary Outcome: Quality of Life Rating Short Form 12-item (SF-12) Health Survey
Description: Assessed by questionnaire rating, compared with pre-intervention rating
  Short form 12-item (SF-12) health survey. Scores range 0%-100%. Score of 0 (minimum) no pain. Score of 100 (maximum) lot of pain. Lower scores is better as it reflect lower pain
Time Frame: Within 1 week of completion of 3-week intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMER | OMT (Osteopathic Manipulative Treatment) | BEMER + OMT | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 46.8 (6.5) | 44.9 (8.9) | 46.0 (11.4) | 48.6 (6.9)

ADVERSE EVENTS:
Time Frame: up to 2 weeks
Arm/Group | BEMER | OMT (Osteopathic Manipulative Treatment) | BEMER + OMT | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04704375/Prot_SAP_002.pdf
  • Informed Consent Form (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04704375/ICF_003.pdf